CLINICAL TRIAL: NCT05132790
Title: Study to Evaluate the Efficacy and Safety of Stereotactic Body Radiation Therapy (SBRT) Combined Neoadjuvant Treatment for Patients With Triple-negative and Hormone Receptor-positive, HER2-negative Breast Cancer
Brief Title: Breast Cancer Study of Stereotactic Body Radiation Therapy (SBRT) Combined Neoadjuvant Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Caigang Liu, professor, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-NEO-IIT-SHR1316-SHR6390-RT
Record Dates: First submitted 2021-11-01; First posted 2021-11-24 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNBC (Experimental)
  Interventions: Drug: SHR-1316 at a dose 20mg/kg q3w; Radiation: SBRT
- HER2-/HR+BC (Experimental)
  Interventions: Drug: SHR6390 at a dose of 150mg orally, daily; Radiation: SBRT

INTERVENTIONS:
Drug: SHR-1316 at a dose 20mg/kg q3w — Combination of SBRT and SHR1316, followed by SHR1316 plus nab-paclitaxel and carboplatin or cisplatin
  Arms: TNBC
Drug: SHR6390 at a dose of 150mg orally, daily — SHR6390 plus exemestane with/without ovarian function suppression/ablation (OFS) after SBRT
  Arms: HER2-/HR+BC
Radiation: SBRT — radiation therapy for breast cance before surgery.

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of stereotactic body radiation therapy (SBRT) combined neoadjuvant treatment for patients with triple-negative and hormone receptor-positive, HER2-negative breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histologic diagnosis of invasive adenocarcinoma of the breast
* ER, PR and HER2 testing, and
* TNBC patients （ HER2-neu 0-1+ by IHC or FISH-negative by ASCO CAP guidelines）
* ER-positive and HER2-negative breast cancer
* tumor measuring ≥2 cm in maximal diameter as measured by any available standard of care imaging (mammogram, breast ultrasound, breast MRI)
* Any nodal status
* ECOG Performance Status of 0 -1
* Screening laboratory values must meet the following criteria:

  i. Absolute neutrophil count (ANC) ≥1.5 × 109/L ii. Platelets ≥100 × 109/L iii. Hemoglobin ≥ 10.0 g/dl for TNBC, ≥ 10.0 g/dl for HR+/HER2-BC iv. Serum creatinine ≤1.5 x upper limit of normal (ULN) v. AST ≤ 2.5 xULN vi. ALT ≤ 2.5 x ULN vii. Total bilirubin ≤ 2.5 xULN viii left ventricular ejection fraction ≥ 50%.

Exclusion Criteria:

* Any kind of prior treatment for breast cancer, including chemotherapy, radiotherapy, endocrine therapy and so on
* Inflammatory breast cancer
* Pregnant and lactating women;
* distant metastasis
* patients who have participated in other clinical trials.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) for TNBC group | Up to11 months
  pCR is defined as the absence of residual invasive cancer on resected breast specimen and the sampled regional lymph nodes as shown by hematoxylin-eosin staining after completion of the neoadjuvant treatment.
Residual cancer burden (RCB) 0-I index for HER2-/HR+BC group | Up to11 months
  Residual cancer burden (RCB) is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. 5 variables are included in a calculation formula to evaluate the total index(0-III), the higher scores mean a worse outcome

SECONDARY OUTCOMES:
Pathological complete response (pCR) forHER2-/HR+BC group | Up to11 months
  pCR is defined as the absence of residual invasive cancer on resected breast specimen and the sampled regional lymph nodes as shown by hematoxylin-eosin staining after completion of the neoadjuvant treatment.
Residual cancer burden (RCB) 0-I index for TNBC group | Up to11 months
  Residual cancer burden (RCB) is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. 5 variables are included in a calculation formula to evaluate the total index(0-III), the higher scores mean a worse outcome

OTHER OUTCOMES:
Objective response rate(ORR) | Up to11 months
  ORR by investigator using RECIST Guideline (Version 1.1)
Adverse reactions（AE） and Serious adverse reactions （SAE) | Through study completion, an average of 15 months
  Adverse reactions（AE） and Serious adverse reactions during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will indicate whether stereotactic body radiation therapy (SBRT) combined neoadjuvant treatment for patients with triple-negative and hormone receptor-positive, HER2-negative breast cancer is safe and effective.

REFERENCES:
- [Derived] Zhang Y, Cao S, Niu N, Shan H, Xue J, Chen G, Xu Y, Yin J, Liu C, Sun L, Jiang X, Tang M, Xu Q, Jia M, Zhang X, Zhang Z, Zhang Q, Wang J, Li A, Yang Y, Liu C. Efficacy and safety of neoadjuvant stereotactic body radiation therapy plus dalpiciclib and exemestane for hormone receptor-positive, HER2-negative breast cancer: A prospective pilot study. Elife. 2025 Jul 28;14:RP101583. doi: 10.7554/eLife.101583. PMID 40719174
- [Derived] Chen G, Gu X, Xue J, Zhang X, Yu X, Zhang Y, Li A, Zhao Y, He G, Tang M, Xing F, Yin J, Bian X, Han Y, Cao S, Liu C, Jiang X, Zhang K, Xia Y, Li H, Niu N, Liu C; Northeastern Clinical Research Alliance of Oncology (NCRAO). Effects of neoadjuvant stereotactic body radiotherapy plus adebrelimab and chemotherapy for triple-negative breast cancer: A pilot study. Elife. 2023 Dec 22;12:e91737. doi: 10.7554/eLife.91737. PMID 38131294